CLINICAL TRIAL: NCT02659007
Title: Less Neuropathy After Yoga
Brief Title: Less Neuropathy After Yoga- Managing Diabetic Neuropathy With Yoga
Acronym: LeNY
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Colorado State University (Other)
Responsible Party: Principal Investigator, Arlene Schmid, Associate Professor, Colorado State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-4894H
Record Dates: First submitted 2016-01-14; First posted 2016-01-20 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Diabetic Neuropathy
Keywords: yoga; balance
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- yoga (Experimental): yoga, 2 times a week for 8 weeks
  Interventions: Other: yoga

INTERVENTIONS:
Other: yoga — 8 weeks of yoga, twice a week. sitting, standing, and floor postures with meditation and breath work

SUMMARY:
The long-term goal is to identify and establish effective mind-body interventions (as an aspect of complementary and alternative medicine) to improve health and Quality of Life (QoL) for people with disabilities. Preliminary data suggest that engagement in yoga is feasible and beneficial for multiple study populations, and it may relieve symptoms of neuropathy. The central hypothesis is that individuals who complete yoga will have significantly better balance, mobility, and QoL after 8 weeks of yoga.

DETAILED DESCRIPTION:
assessments completed before and after yoga. yoga was delivered twice a week for 8 weeks for one hour each session. Yoga included sitting, standing, and floor postures, breath work, and meditation

ELIGIBILITY:
Inclusion Criteria:

* Anyone age 18 and over with DPN from Diabetes Mellitus and a balance impairment. and be able and willing to attend twice weekly sessions for 8 weeks.

Exclusion Criteria:

* not have consistently engaged in yoga for greater than a year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
change in Neuro-QoL | baseline and 8 weeks
  used to assess health related quality of life in people with neuro disability
change in Berg balance Scale | baseline and 8 weeks
  assess static and dynamic balance
change in 6 minute walk | baseline and 8 weeks
  amount of feet walked in 6 minutes, used to assess endurance
change in 10 meter walk | baseline and 8 weeks
  amount of time to walk 10 meters, measures gait speed

IPD SHARING:
Plan to Share IPD: No